CLINICAL TRIAL: NCT04556344
Title: Effectiveness of an Educational Intervention Aimed at Increasing the Emotional Competencies of Patients Under Surveillance After Antineoplastic Treatment of Oesogastric or Bronchopulmonary Cancer: a Randomized, Multicenter, Controlled Pilot Study (EmoVie-K2)
Brief Title: Effectiveness of an Educational Intervention Aimed at Increasing the Emotional Competencies of Patients Under Surveillance After Antineoplastic Treatment of Oesogastric or Bronchopulmonary Cancer
Acronym: EmoVie_K2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: SCALab UMR CNRS 9193 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019_69; 2020-A00674-35 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2020-09-08; First posted 2020-09-21 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2022-05

CONDITIONS: Digestive System Neoplasms; Thoracic Neoplasms
Keywords: Emotional Intelligence; Quality of Life; cancer survivors; psychology; supportive care
MeSH Terms: conditions — Digestive System Neoplasms; Thoracic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional skills (Experimental): 3 individual sessions in which patients are going to learn how to identify, understand, express and regulate emotions
  Interventions: Behavioral: Emotional skills
- Short free talk and relaxation (Sham Comparator): 3 individual sessions in which patients are going to follow relaxation instructions after a non-directive talk about their current or past experience of cancer.
  Interventions: Behavioral: Short free talk and relaxation

INTERVENTIONS:
Behavioral: Emotional skills — 3 sessions of 1,5 hour each. The first session can be face to face or over the phone, the two last ones will be held over the phone.
  Arms: Emotional skills
Behavioral: Short free talk and relaxation — 3 sessions of 1,5 hour each. The first session can be face to face or over the phone, the two last ones will be held over the phone.
  Arms: Short free talk and relaxation

SUMMARY:
Emotional skills are the ability to use emotions cleverly in daily life. Good emotional skills are associated with better mental and physical health in healthy and clinical populations. However, to our knowledge, cancer patients have never benefited from an intervention aiming at increasing their emotional skills. Our goal was thus to design and test such an intervention. A prospective, multi-center, randomized controlled trial (RCT) will be conducted in esogastric and lung cancer patients after antineoplastic treatments. Forty-three patients are expected in each arm. The primary outcome is the change in emotional skills assessed using a patient-reported validated questionnaire between the start and two weeks after the end of the intervention and at 2-month follow-up. The experimental arm will have to follow three individual sessions on emotional skills (i.e. identification, understanding, expression and regulation of emotions) while the control arm will have to follow three sessions of relaxation. In each arm, the first session can be held face to face or over the phone and the last two sessions will be held over the phone. Patients have exercises to practice in between sessions.It is hypothesised that the experimental group will experience a greater increase in emotional skills than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patient under surveillance after curative or palliative antineoplastic treatment (surgery and/or chemoradiotherapy and/or radiotherapy alone and/or chemotherapy alone) of esogastric or bronchopulmonary cancer,
* Patients with a life expectancy estimated by their physician involved in the research to be greater than or equal to six months,
* Patient with a ≥ 4 score on the Distress Scale (scale from 0 to 10),
* Affiliation to a social security scheme,
* Mastery of the French language,
* Signing of informed consent to participate in this research.

Exclusion Criteria:

* Cognitive disorders or unstabilized psychiatric disorders that may impair the ability of reasoning and thinking necessary to complete the questionnaires and attend workshops
* Difficulty or deficiency that prevent the patient from a good understanding of the imperatives of the research
* Any situation likely to significantly affect emotional competence during the study according to the investigator's judgment (in particular, ongoing psychotherapeutic follow-up))
* Patients under judicial protection (guardianship or curators).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Change in patient emotional skills from baseline to 15 days after the end of intervention | Between Baseline (T0) and 15 days after the intervention (T1)
  Variation in patient-reported 13-item Short Profile of Emotional Competence (S-PEC) score from baseline (T0) to 15 days after the intervention (T1)

SECONDARY OUTCOMES:
Patient emotional skills at follow up | Between T0 (start of the intervention) and T2 (2 months after T1)
  Variation in the emotional competence score (13-item S-PEC) between Baseline (T0) and T2 (2.5 months after the last session).
Difficulties in Emotional Regulation | Between T0 (baseline) and T1 (15 days after the end of the intervention) and between T1 and T2 (2 months after T1)
  Variation in the Difficulties in Emotional Regulation Scale (DERS 16) score between T0 and T1 and between T1 and T2.
Quality of life by FACT-G | At T0 (before the first session), at T1 (15 days after the last session) and at T2 (2 months after T1).
  Patients' self-reported quality of life assessed using the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire
Change in quality of life using FACT-G | Between T0 (baseline) and T1 (&5 days after the end of the intervention) and between T1 and T2 (2 months after T1)
  Variation in assessed quality of life (FACT-G) between T0 and T1 and between T1 and T2 based on variation in emotional competence (13-item S-PEC)
Patient participation in workshops | Between 2 weeks and 2 months
  The percentage of patients who have attended the 3 group sessions
Patient adherence to exercises to do at home between sessions | Between 2 weeks and 2 months
  The percentage of patients who have performed the suggested exercises at home between sessions
Patient satisfaction | T1 (15 days after the end of the intervention) and T2 (2 months after T1)
  Patient-reported satisfaction regarding the intervention using ad hoc questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Cortot, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Calmette,CHU, Lille, France